CLINICAL TRIAL: NCT06215066
Title: Effect of Virtual Reality and Modified Progressive Muscle Relaxation Distraction Techniques on Anxiety and Attention Among Cardiac Care Unit Patients; RCT.
Brief Title: Effect of Virtual Reality and Progressive Muscle Relaxation on Anxiety and Attention Among Cardiac Care Unit Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Collaborators: Middle East University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Distraction Techniques
Record Dates: First submitted 2023-09-21; First posted 2024-01-22 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Anxiety
Keywords: Anxiety, Attention, Distraction Techniques, MPMR, VR.
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A total sample of 158 patients was required. A computer randomizer (www.randomizer.org
  ) was used to assign numbers to patients who were included. A 1:1 randomized allocation was applied to assign patients to each group. As an active comparator, Group A received the virtual reality (VR) intervention (83 patients), whereas Group B received the modified progressive muscle relaxation (MPMR) intervention (75 patients). Blinding in this study was limited to the statistician.
Who Masked: Outcomes Assessor
Masking Description: Blinding was limited to the statistician (outcome assessor). Participants, care providers, and investigators were not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Group (VR) (Active Comparator): The intervention was administered three times per day, 10 minutes each session, for three consecutive days.
  The VR goggles and headset phone were placed on the patient's head, straps secured, and lens spacing adjusted for a clear visual field. Patients were instructed to use head movements to control the cursor and interact with the virtual content. The 3D video clips with natural sceneries and background music were played to create a relaxing experience.
  Interventions: Device: Virtual reality
- Modified Progressive Muscle Relaxation Group (MPMR) (Active Comparator): The intervention was administered three times per day, 10 minutes each session, for three consecutive days.
  The exercises applied to specific body parts while patients closed their eyes and practiced deep breathing, accompanied by background music.
  Interventions: Other: Modified Progressive Muscle Relaxation

INTERVENTIONS:
Device: Virtual reality — The VR goggles and headset phone were placed on the patient's head, straps secured, and lens spacing adjusted for a clear visual field. Patients were instructed to use head movements to control the cursor and interact with the virtual content. The 3D video clips with natural sceneries and background music were played to create a relaxing experience.
  Other Names: VR
  Arms: Virtual Reality Group (VR)
Other: Modified Progressive Muscle Relaxation — The exercises applied to specific body parts while patients closed their eyes and practiced deep breathing, accompanied by background music.
  Other Names: MPMR
  Arms: Modified Progressive Muscle Relaxation Group (MPMR)

SUMMARY:
A randomized controlled trial with two parallel groups was conducted, to determine the effect of virtual reality (VR) and modified progressive muscle relaxation (MPMR) distraction techniques on anxiety, attention and getting distracted from the external environment among cardiac care unit patients.

The study is based on the following hypotheses:

H1: Patients who receive VR intervention have lower Hamilton Anxiety Rating (HAM-A) scores than those who receive MPMR intervention.

H2: Patients who receive VR intervention exhibit improvement in their physiological parameters than those who receive MPMR intervention.

H3: Patients who receive VR intervention have higher Attention/Distraction scores than those who receive MPMR intervention.

DETAILED DESCRIPTION:
This randomized controlled trial with two parallel groups was conducted in the cardiac care unit of Smouha Hospital, affiliated with Alexandria University, Egypt.

A total of 158 patients were recruited using a simple random sampling method and assigned to one of two groups to determine the effects of virtual reality (VR) and modified progressive muscle relaxation (MPMR) distraction techniques on anxiety, attention, and distraction from the external environment among cardiac care unit patients.

Four assessment tools were used:

1. Sociodemographic and Clinical Assessment.
2. Physiological Parameter Assessment.
3. Hamilton Anxiety Rating Scale (HAM-A).
4. Attention/Distraction Scale.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to CCU for at least 3 days after stability.
* Patients who are conscious and stable condition and all of whom exhibited varying levels of anxiety.

Exclusion Criteria:

- Patients with a history of neurological impairments such as motor, visual, and auditory disabilities and psychological disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-24 (Actual)

PRIMARY OUTCOMES:
Comparison of changes in physiological parameters between baseline and post-intervention scores for both groups. | Baseline physiological parameter assessments were conducted individually for each patient on the first day of the intervention. Post-intervention assessments were conducted during the same three shifts across the three-day period.
  Compares the degree of change between baseline physiological parameters (heart rate and rhythm, respiratory rate and rhythm, oxygen saturation, blood pressure, and pain level) and post-intervention scores for both groups.

SECONDARY OUTCOMES:
Comparison of changes in anxiety levels between baseline and post-intervention scores for both groups. | Baseline anxiety level assessments were conducted individually for each patient on the first day of the intervention. Post-intervention assessments were conducted during the same three shifts across the three-day period.
  Compares the degree of change between baseline anxiety level (Hamilton Anxiety Rating Scale, HAM-A) and post-intervention scores for both groups.

OTHER OUTCOMES:
Comparison of attention / distraction levels between both groups at the end of the intervention. | Attention / distraction levels were assessed individually for each patient during the night shift on the third day after completing all nine intervention sessions.
  Compares attention / distraction levels using the Attention / Distraction Scale for both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Sajeda A Shdaifat, PhD-Cand, Principal Investigator — Alexandria University; Azza H El-Soussi, Professor, Study Director — Alexandria University; Mohamed I Sanhoury, Asst. Prof, Study Director — Alexandria University; Eman A Ali, Asst. Prof, Study Director — Alexandria University
Locations (1):
- Cardiac care unit of Smouha Hospital, which is affiliated to Alexandria University, Egypt., Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No